CLINICAL TRIAL: NCT03992001
Title: Prospective Crossover Study on Beta(ß)-Thalassaemia Transfusion-dependent to Evaluate the Impact on Transfusion Regimen of Two Pre-storage Leukoreduced PRBCs(In-line Filtration + B-C Separation; Whole Blood Filtration + B-C Conservation)
Brief Title: Impact of the Preparation Method of Red Cell Concentrates on Transfusion Indices in Thalassemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Maria Rita Gamberini, Head, Day Hospital Thalassaemia and Haemoglobinopathies (DHTE) - Azienda Ospedaliero-Universitaria S.Anna of Ferrara, Università degli Studi di Ferrara
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CrossoverFE2018
Record Dates: First submitted 2018-11-15; First posted 2019-06-19 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Thalassemia Major
Keywords: Packed RBCs; leukodepletion; buffy-coat; transfusion
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups of approximately equal number. The first group will receive the blood component A for a period of 6 months and then the blood component B for the next 6 months. The second group will receive the blood components in inverted order
Masking Description: The patients will not be informed on the blood components sequence that they will receive. However, the units exterior appearance of the two types of preparations is different. For this reason, patients and care providers will most probably notice it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A-B (Experimental): Patients in this arm will receive blood component A for 6 months and blood component B for the next 6 months
  Interventions: Biological: Blood component A; Biological: Blood component B
- Sequence B-A (Experimental): Patients in this arm will receive blood component B for 6 months and blood component A for the next 6 months
  Interventions: Biological: Blood component A; Biological: Blood component B

INTERVENTIONS:
Biological: Blood component A — PRBCs obtained from whole blood after separation of plasma, buffy coat, and RBCs and successive leukoreduction of RBCs
Biological: Blood component B — PRBCs obtained by leukoreduction of whole blood, and successive separation of plasma and RBCs

SUMMARY:
This study compares the effects of Packed Red Blood Cells (PRBCs) prepared in two different ways on the transfusion indices in beta(ß)-Thalassemia transfusion-dependent patients. The two blood components types derive from the whole blood. In one case, the whole blood is leukoreduced with subsequent plasma removal. In the other case, plasma, buffy coat, and red blood cells (RBCs) are first separated and subsequently, the RBCs leukoreduced. Each type of blood components will be subsequently given to one-half of the patients for a 6-month period and to the other half for other 6-month at the randomization phase, for a total of 12 months of crossed-treatment per patient.

DETAILED DESCRIPTION:
At Day Hospital Talassemia ed Emoglobinopatie of Ferrara, two different PRBCs are available. The two types of blood components are obtained from whole blood, pre-storage leukoreduced and suspended in saline-adenine-glucose-mannitol (SAGM). One method of preparation consists of the whole blood leukoreduction with subsequent plasma removal. The other method first separates plasma, buffy coat, and RBCs, and then the RBCs are leukoreduced. The two methods mainly differ in the final haemoglobin (Hb) content: the Hb level is lower (-13%, approximately) in the second method that also shows the advantage to produce platelets from the buffy coat. A PRBCs unit is not as strictly defined as a therapeutic medication dose (pill or vial): individual PRBCs units may substantially differ in their Hb content, much more than the average difference between the two types of preparations. The aim of this study is to document the extent of the average difference between the two types of preparations, and its impacts on the transfusion indices of ß-Thalassaemia transfusion-dependent patients. All patients will receive each blood component for a period of 6 months (crossover design), for a total of 12 months of transfusion treatment per patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient with beta(ß)-Thalassaemia transfusion-dependent (ß-Thalassemia Major or ß-Thalassemia Intermedia transfusion-dependent, regularly transfused since at least 5 years

Exclusion Criteria:

* Patient not exclusively transfused at Day Hospital Thalassaemia and Haemoglobinopathies of Ferrara
* Patient with haemolytic auto-antibodies
* Patient transfused with washed Packet RBCs units
* Severe splenomegaly (>18 cm on echography)
* Elevated blood consumption (>200 mL/kg of pure RBCs in the last year)
* Patient receiving haemoglobin inducers in the last 6 months
* Any significant clinical pulmonary, cardiovascular, endocrine, hepatic, gastrointestinal, renal, infectious, immunological including significant allo- or auto-immunisation disease, considered not adequately controlled prior to the study
* Patient treated with erythrocyte exchange
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Transfusion Power Index | For each of the two blood components studied, at the end of 6-month period of study
  (Average pre-transfusion Hb concentration)/(Unit Index) [for the definition of Unit Index, see the secondary outcomes]

SECONDARY OUTCOMES:
Average pre-transfusion Hb concentration | For each of the two blood components studied, at the end of 6-month period of study
  Mean pre-transfusion Hb levels, calculated starting from the second transfusion of the period to the first transfusion of the following period
Unit Index | For each of the two blood components studied, at the end of 6-month period of study
  (Total number of PRBCs (A or B) transfused in the period)/(Number of days between the first transfusion of the period and the first transfusion of the following period)
Average Transfusion Interval | For each of the two blood components studied, at the end of 6-month period of study
  (Number of days between the first transfusion of the period and the first transfusion of the following period)/(Number of transfusions in the period)
Number of Transfusion Reactions | Study periods (2 periods of 6 months each)
  Number of transfusion reactions to the two blood components that may occur in the study periods (2 periods of 6 months each)
Transfusion Reaction Rate | Study periods (2 periods of 6 months each)
  (Number of transfusion reactions to the two blood components occurring in the study periods)/(Total number of PRBCs (A or B) transfused in the period)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rita Gamberini, MD, Study Chair — D.H. Thalassaemia-Haemoglobinopathies (DHTE) - A.O.U. S. Anna of Ferrara
Locations (1):
- Day Hospital Thalassaemia and Haemoglobinopathies (DHTE), Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD (deidentified) available to other researchers and support already published results
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication
Access Criteria: Please contact the Central Contact Person